CLINICAL TRIAL: NCT07066007
Title: First Aid Training Booklet for Parents of Children 0-6 Years Old
Brief Title: Evaluation of the Effectiveness of the First Aid Program Applied to Parents of 0-6 Year Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semra SÖNGÜT (Other)
Responsible Party: Sponsor-Investigator, Semra SÖNGÜT, Lecturer, Hitit University
Organization: Hitit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-12
Record Dates: First submitted 2025-05-23; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Increasing the First Aid Knowledge and Practice Levels of Parents; Accidental Injuries; Pediatric Emergency Care; First Aid Training; Child Safety; Self Efficacy
Keywords: 0-6 years old child; Parent education; Education program; First aid
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group will not be distributed to education
- First Aid Education Program for Parents (Experimental): Parents of 0-6-year-old children who received a structured first aid education program consisting of 6 modules over 3 sessions (each session 120 minutes), including theoretical instruction, hands-on practice, and case simulations. Topics include pediatric emergencies, trauma management, and self-efficacy development.
  Interventions: Behavioral: First Aid Education Programme

INTERVENTIONS:
Behavioral: First Aid Education Programme — A six-module behavioral education program for parents, designed to improve first aid knowledge, application skills, and self-efficacy. Delivered face-to-face in three 120-minute sessions using theoretical lectures, demonstrations, and case-based simulations.
  Arms: First Aid Education Program for Parents

SUMMARY:
Purpose: Accidents/injuries seen in children aged 0-6 in developed and developing countries are among the leading preventable health problems and are among the leading causes of death and disability. In the event of an accident/injury, many children can be saved and/or complications can be prevented with correct first aid knowledge and practices until the health team arrives. Therefore, parents are the first to have first aid knowledge and skills, and first aid training given to parents is very important so that they can provide correct first aid intervention in the event of an accident/injury. In this way, it will be possible to increase parents' awareness and self-efficacy, and mortality and morbidity rates after accidents/injuries in children can be reduced. It is important for pediatric nurses, who are important members of preventive health services, to create educational content according to the target audience and to provide first aid training to parents accordingly. In this context, the aim of this study is to evaluate the effectiveness of the first aid training program given to parents of 0-6 year old children, to improve parents' first aid application skills and to increase their first aid self-efficacy levels.

Scope and Objectives: In this project covering parents of 0-6 year old children; it is aimed to increase parents' first aid knowledge level, application skills and first aid self-efficacy.

Method: This study is planned as a randomized controlled experimental study. Parents of 0-6 year old children registered in Çorum Province Family Health Centers and nurseries and kindergartens affiliated with the Ministry of Family and Social Policies will be included in the study group. The parents participating in the study will be randomized into intervention and control groups. Parents will be divided into strata according to their level of education and the ages of their children, and stratification will be carried out after the pre-test of the study is applied. Parents will not be informed whether they are in the intervention or control group. The intervention group will be trained with the "First Aid Training Booklet for Parents of 0-6 Year Old Children" developed by the researchers. After the training, a post-test will be applied to the intervention and control groups. The research data will be collected using the "Introductory Information Form", "First Aid Knowledge Evaluation Form", "First Aid Application Skill Evaluation Form" and "First Aid-Self-Efficacy Scale" through face-to-face interviews.

Expected Results: The training program prepared for parents of children aged 0-6;

* It can be used in all scientific studies such as research, thesis, and projects planned to be conducted in the field,
* It can be used as a resource if "first aid" courses are added to the postgraduate education curricula of "Pediatric Nursing", "Public Health Nursing", "Surgical Diseases Nursing", which are frequently in contact with children of this age,
* It can form the basis for projects planned within the scope of "training of trainers" for students receiving postgraduate education in the fields of "Pediatric Nursing", "Public Health Nursing", "Surgical Diseases Nursing",
* Proper and effective first aid applications allow children to continue their lives in a healthy way by providing timely intervention. It is thought that the health of children, who are the future of societies, will contribute to the reduction of the frequency of applications for treatment and care services at health institutions and, in this respect, the effective use of economic resources allocated by governments to health.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children between the ages of 0-6,
* Parents who can read and write in Turkish,
* Parents who volunteer to participate in the research.

Exclusion Criteria:

* Parents who have received first aid training in the last 3 years,
* Parents who have not completed first aid training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
First Aid Knowledge Score | Baseline (Day 0) and immediately after intervention (Week 2)
  The 101-question "First Aid Knowledge Evaluation Form" developed by the researcher is used to assess parents' knowledge of pediatric first aid. Scores range from 0 to 101; higher scores indicate higher knowledge levels.
  The form is grouped according to the modules in the training program. In this context, it consists of a total of 101 questions: Module 1: General First Aid Information (14 questions); Module 2: Basic Life Support (BLS) Information (16 questions); Module 3: First Aid Information in Traumatic Injuries (31 questions); Module 4: First Aid Information in Medical Emergencies (18 questions); Module 5: First Aid Information in Other Emergencies (22 questions). Each question on the form was evaluated with two options as "true" and "false". It was scored as "Correct answers = 1" and "Wrong answers = 0". Accordingly, the total score that each parent can get from the "First Aid Knowledge Evaluation Form" was evaluated between 0 and 101.

SECONDARY OUTCOMES:
First Aid Practice Score | Baseline (Day 0) and immediately after intervention (Week 2)
  The 100-question "First Aid Application Skills Evaluation Form" developed by the researcher is used to evaluate parents' application skills in pediatric first aid. Observational checklist used to evaluate parents' first aid application skills. Structured performance checklist includes critical steps in pediatric emergencies. Scores range from 0 to 101; higher scores reflect better skill performance.The form is grouped according to the modules in the training program. In this context, it consists of a total of 100 questions: Module 1: Basic First Aid Application Skills (14 questions); Module 2: Basic Life Support (BLS) Application Skills (9 questions); Module 3: First Aid Application Skills in Traumatic Injuries (39 questions); Module 4: First Aid Application Skills in Medical Emergencies (18 questions); Module 5: First Aid Application Skills in Other Emergencies (20 questions). Each question on the form was evaluated with two options as "applied" and "could not apply".

OTHER OUTCOMES:
First Aid Self-Efficacy Score | Baseline (Day 0) and immediately after intervention (Week 2)
  First Aid-Self-Efficacy Scale was developed by Gülmez Dağ and Çapa Aydın (2015) in order to assess how competent individuals feel in first aid applications. This scale, developed as a nine-point Likert-type scale, consists of a total of 25 items. These items are scored as "1: insufficient; 2-3: very competent; 4-5: somewhat competent; 6-7: quite competent; 8-9: very competent". While items 2, 8, 10, 14, 17, 18, 19 and 20 of the scale cover the knowledge dimension of "Life Support First Aid Self-Efficacy", items 1, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 16, 21, 22,23, 24 and 25 cover the skill and competence dimension of "Basic First Aid Self-Efficacy". As a result of the reliability analysis of the scale, Cronbach's Alpha coefficient was determined as 0.96 for the first dimension and 0.91 for the second dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)